CLINICAL TRIAL: NCT05125900
Title: Clinical Evaluation of Subgingival Open Sandwich Restorations: 3-year Results of a Randomized Double-blind Trial
Brief Title: Clinical Evaluation of Subgingival Open Sandwich Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A01111219
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Dental Restoration Failure of Marginal Integrity
Keywords: Deep margin elevation; Proximal box elevation; Open sandwich technique; Bi-layered restorations; Subgingival cervical margin

STUDY DESIGN:
Intervention Model Description: Each patient received one or two restorations in a posterior tooth on any side randomly selected from the 4 tested restorative materials, all materials were used according to manufacturers' instructions
Who Masked: Participant, Investigator
Masking Description: Double (Participant and Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Resin modified glass ionomer (Active Comparator): Group received proximal box elevation using resin modified glass ionomer
  Interventions: Other: Proximal box elevation using one of the tested materials
- Glass hybrid (Placebo Comparator): Group received proximal box elevation using glass hybrid
  Interventions: Other: Proximal box elevation using one of the tested materials
- Bulk fill flowable resin composite (Active Comparator): Group received proximal box elevation using bulk fill flowable resin composite
  Interventions: Other: Proximal box elevation using one of the tested materials
- Ion-releasing material (Placebo Comparator): Group received proximal box elevation using ion-releasing material
  Interventions: Other: Proximal box elevation using one of the tested materials

INTERVENTIONS:
Other: Proximal box elevation using one of the tested materials — Each patient randomly received deep proximal margin elevation with one of the tested restorative materials, while the overlying restorations were all the same regular bulk fill resin composite

SUMMARY:
This study was designed to evaluate and compare the 3-year periodontal responses and clinical performance of proximal subgingival open sandwich restorations using three different glass ionomer-based restorative materials and flowable composite.

DETAILED DESCRIPTION:
The description of the experimental design followed the Consolidated Standards of Reporting Trials (CONSORT) statement. The present study was a double-blinded (patients and examiner) randomized clinical trial anticipating the parallel design. Ninety-five adult patients seeking dental treatment in the Operative Department clinic at the Faculty of Dentistry, University of Mansoura were enrolled in the current study with a total of 120 Class II restorations. No advertisement was made for participant recruitment, forming a sample of convenience. Each patient must signs a consent form before participating in the current study. The study was conducted from January 2020 to January 2023 as a part of the Doctoral dissertation. Mansoura University institution's ethics committee approved the form and protocol before conducting the study. The sample size was calculated based on the clinical success rate (100% success rate at 2 years) of posterior class II restorations restored with open sandwich and deep margin elevation techniques observed in previous studies. According to several parameters including a significance level of 5%, the power of the test was calculated to be 80%, and equivalent limit of 15%. Upon these data, a sample size of 120 subjects was appropriate to allow for a 20% drop-out.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one proximal sub gingival carious lesion ICDAS 4, or 5 in posterior teeth
* Patients must have a good oral hygiene;
* Patients with tooth gives positive response to testing with an electric pulp tester
* Patients with normal and full occlusion,
* Patients with opposing teeth should be natural with no restorations.

Exclusion Criteria:

* High caries risk patients with extremely poor oral hygiene,
* Patients involved in orthodontic treatment or periodontal surgery,
* Patients with periodontally involved teeth (chronic periodontitis)
* Patients with abutments should be excluded.
* Patients with heavy bruxism habits and clenching

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with periodontal problems | 3 years after restoration
  The periodontal situation of patients were examined based on bleeding on probing, plaque index and probing depth scores
Percentage of aesthetic, functional and biological properties for each base material restorations | 3 years after restoration
  Percentage of aesthetic, functional and biological properties were clinically assessed using World Dental Federation parameters for each base material group

SECONDARY OUTCOMES:
Radiographic examination | 3 years after restoration
  Each base material/gingival dentin interface was examined radiographically each 6 months period.

CONTACTS AND LOCATIONS:
Overall Officials: Hoda S Ismail, Lecturer, Principal Investigator — Faculty of Dentistry, Mansoura University, Egypt
Locations (1):
- Faculty of Dentistry-Mansoura University, Al Mansurah, Dakahliya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Statistical Analysis Plan can be shared to other researchers
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available within 6 Months for 3 years
Access Criteria: for anyone